CLINICAL TRIAL: NCT02587611
Title: Randomized Comparison of Elemental Liquid Diet and Standard Semi-solid Diet on Gastric Emptying in Healthy Subjects and Bedridden Gastrostomy-fed Patients
Brief Title: Randomized Comparison of Elemental Liquid Diet and Standard Semi-solid Diet on Gastric Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Showa Inan General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Gastric emptying
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Gastric Emptying

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elemental liquid diet (Experimental): Elemental liquid diet (200 kcal/200 mL) is labeled with 100 mg [13C]sodium acetate and healthy subjects drink it within 5 min.
  Elemental liquid diet (200 kcal/200 mL) is labeled with 100 mg [13C]sodium acetate and is administered within 15 min using the gastrostomy tube.
  Interventions: Other: Elemental liquid diet
- Standard semi-solid diet (Active Comparator): Standard semi-solid diet (200 kcal/200 mL) is labeled with 100 mg [13C]sodium acetate and healthy subjects drink it within 5 min.
  Standard semi-solid diet (200 kcal/200 mL) is labeled with 100 mg [13C]sodium acetate and is administered within 15 min using the gastrostomy tube.
  Interventions: Other: Standard semi-solid diet

INTERVENTIONS:
Other: Elemental liquid diet — This is a randomized, crossover trial. Two types of test meals (200 kcal/200 mL of either the elemental diet or the semi-solid diet) are labeled with 100 mg [13C]sodium acetate and administered within 5 min in healthy subjects or within 15 min in gastrostomy-fed patients.
  Other Names: Elental®
  Arms: Elemental liquid diet
Other: Standard semi-solid diet — This is a randomized, crossover trial. Two types of test meals (200 kcal/200 mL of either the elemental diet or the semi-solid diet) are labeled with 100 mg [13C]sodium acetate and administered within 5 min in healthy subjects or within 15 min in gastrostomy-fed patients.
  Other Names: Racol NF semi-liquid®
  Arms: Standard semi-solid diet

SUMMARY:
The purpose of this study is to compare the effect of either elemental liquid diet or standard semi-solid diet on gastric emptying in both healthy subjects and bedridden patients receiving gastrostomy feeding.

DETAILED DESCRIPTION:
A randomized, crossover trial using elemental liquid diet or standard semi-solid diet containing 13C sodium acetate as a tracer is performed in both healthy subjects and bedridden gastrostomy-fed patients. 13C breath tests is performed to estimate gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects bedridden gastrostomy-fed patients

Exclusion Criteria:

* regular use of gastric acid blockers, motility drugs, benzodiazepines or opioids, any clinical evidence of acute infection, a history of abdominal surgery, and an American Society of Anesthesiologists physical status of class IV or V.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 4 hours
  10% 30% or 50% gastric emptying (excretion) time

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, MD, Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General Hospital, Komagane, Japan